CLINICAL TRIAL: NCT01865240
Title: Renal Denervation for Resistant Hypertension
Acronym: RDNP-2012-01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No new participants enrolled. Protocol has been superseded
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008/12; NHMRC (Other Grant/Funding Number: 1034397)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Hypertension
Keywords: renal denervation; blood pressure; cardiovascular risk; target organ damage; sympathetic activity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Denervation Group (Experimental): participants randomised to undergo the renal denervation procedure
  Interventions: Device: Renal Denervation
- Usual care (No Intervention): participants randomised to the usual care group will receive additional antihypertensive medication in an attempt to achieve blood pressure targets

INTERVENTIONS:
Device: Renal Denervation — Renal Denervation Catheter
  Other Names: Symplicity Renal Denervation Catheter
  Arms: Renal Denervation Group

SUMMARY:
This is a study investigating the effectiveness of renal denervation in lowering blood pressure in people whose blood pressure is not adequately controlled despite treatment with 3 or more blood pressure lowering drugs. The study is designed to compare the effects of renal denervation to a usual care group receiving additional blood pressure lowering drugs.

DETAILED DESCRIPTION:
Previous studies have shown that the renal denervation procedure is safe and effective in reducing blood pressure in patients with resistant hypertension. A total of 100 participants with uncontrolled blood pressure, treated with three or more blood pressure lowering medications will be recruited into the study. Patients will be assigned to one (1) of two (2) groups with the aim of attaining blood pressure control. Participants in group 1 will be assigned to renal denervation, participants in group 2 will receive additional antihypertensive medication according to current guidelines and best practice in an attempt to reach blood pressure targets.

ELIGIBILITY:
Inclusion Criteria:

* systolic BP ≥140mmHg or ≥130mmHg for patients with diabetes
* concurrent treatment with ≥3 anti-hypertensive drugs

Exclusion Criteria:

* renal artery anatomy ineligible for treatment
* eGFR <15mL/min/1.73m2 (using Modification of Diet in Renal Disease (MDRD) calculation)
* female participants of childbearing potential must have negative pregnancy test prior to treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
blood pressure control | 6 months post procedure
  percentage of patients to achieve Blood Pressure (BP) target (BP <140/90mmHg, or <130/80mmHg in diabetic patients) at 6 months post procedure

SECONDARY OUTCOMES:
number of drugs required to reach blood pressure target | baseline to 6 months
  number of drugs required to reach blood pressure target
time to achieve blood pressure target | baseline to 6 months
  time to achieve blood pressure target
Change in markers of sympathetic nerve activity | baseline to 6 months
  Changes in Muscle Sympathetic Nerve Activity (MSNA), renal and whole body Norepinephrine (NE) spillover
Change in Left Ventricular Structure and Function | baseline to 6 months
  Change in Left Ventricular mass index, ejection fraction, diastolic filling as assessed by echocardiogram
Change in Quality of Life | baseline to 6 months
  Change in Quality of Life as assessed by relevant questionnaires
Serum and Urine Biochemistry | baseline to 6 months
  Plasma renin activity, aldosterone, estimated Glomerular Filtration Rate (eGFR), urine albumin-to-creatinine ratio (UACR), inflammatory markers, 24hour urinary creatinine clearance, sodium, fasting glucose, fasting insulin, c-peptide, Homeostasis Model Assessment (HOMA) index, lipid profile
Change in markers of arterial stiffness | baseline to 6 months
  Change in markers of arterial stiffness including Augmentation Index (AI) and Pulse Wave Velocity (PWV)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, MD, Principal Investigator — Baker IDI Heart & Diabetes Institute
Locations (1):
- Baker IDI Heart & Diabetes Inst, Melbourne, Victoria, Australia